CLINICAL TRIAL: NCT04999033
Title: The Development of Patient Experience With Nursing Care Scale in China
Brief Title: The Development of Patient Experience With Nursing Care Scale
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: B2020-074R
Record Dates: First submitted 2021-08-08; First posted 2021-08-10 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Patient Experience; Nurse-Patient Relations
Keywords: patient experience; nursing care; scale

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Inpatient: This study is a cross-sectional study and no intervention will be involved
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — This is a cross-sectional study, and no intervention will be included

SUMMARY:
Nurses are a vital and central part of the health care system, accounting for nearly half of the global health workforce and spending more time with patients than any other medical professionals. Patient experience with nursing care, as a process indicator, reflects the interpersonal aspects of care received and has an important impact on overall experience and satisfaction with hospital care. The results of the previous study showed that the most important predictor of patient satisfaction with hospitals was patient experiences with nursing care.

Since nurses are so deeply and widely involved in patients' care, an instrument with a clear conception definition, systematically developed and psychometrically validated will be extremely valuable in measuring patient experience with nursing care, so as to collect and analyze patient feedback toward nursing services, and push the quality improvement according to the preferences, needs and values of the healthcare recipients.

This study, therefore, aimed to develop construct and validate a comprehensive and internally consistent instrument to measure patient experience with nursing care in the Chinese hospital setting.

ELIGIBILITY:
Inclusion Criteria:

1. had been hospitalized for 2 days or more;
2. able to speak and understand Chinese.

Exclusion Criteria:

patients with cognitive impairment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible inpatients will be invited to participate the study. For anonymity, participants will be are identified with the letter P followed by a number
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-08 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
patient experience with nursing care | September. 2021
  how often patient experience with each nursing service by using a Likert-type scale ranging from 1 (never) to 5 (always). For each item, the patients will be offered the option of indicating whether it is not relevant.

SECONDARY OUTCOMES:
patient satisfaction with nursing care | September. 2021
  patients will be asked one more questions regarding their satisfaction toward nursing care 'All in all, are you satisfied with the nursing care you received at the hospital?', with a ten-point response option ranging from 1-10 (with 1 labeled "not at all satisfied" and 10 labeled "to a very large extent satisfied").

CONTACTS AND LOCATIONS:
Locations (1):
- 180 Fenglin Road, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
We will share sociodemographic characteristics (For anonymity, participants are identified with the letter P followed by a number) and patient experience data of patients to other researchers when asked
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code